CLINICAL TRIAL: NCT02782533
Title: DBS of the Third Ventricle for Cluster Headache and Obesity
Acronym: DBS V3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU Grenoble
Record Dates: First submitted 2016-05-12; First posted 2016-05-25 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2018-07

CONDITIONS: Cluster Headache; Obesity
MeSH Terms: conditions — Cluster Headache; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DBS V3 (Experimental): Deep Brain Stimulation V3
  Interventions: Device: Deep Brain Stimulation V3

INTERVENTIONS:
Device: Deep Brain Stimulation V3

SUMMARY:
Study of Deep Brain Stimulation of the Third ventricle in Cluster Headache and Obesity treatment.

ELIGIBILITY:
Inclusion Criteria :

* Male or female aged between 18 and 65 years
* Ambulatory or hospitalized monitoring
* Fluent in French and able to understand the study procedures, including completing the auto-questionnaires
* Registered in the French social security scheme
* Signed informed consent of the patient will be collected before inclusion in the study
* Cluster Headache or Obesity patients

Exclusion Criteria:

* Contraindication to Magnetoencephalography (MEG) and/or Electroencephalography (EEG)
* Contraindication to Magnetic resonance imaging (MRI)
* All categories of protected persons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-11; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life Questionnaire | weekly up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- CLINATEC, Grenoble, France

IPD SHARING:
Plan to Share IPD: No